CLINICAL TRIAL: NCT03927989
Title: Tobacco Treatment in the Context of Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00068951
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Advice to quit and brief discussion of tobacco use plus dual nicotine replacement therapy plus 8 weeks of gain-framed text messages tailored to lung cancer screening patients
  Interventions: Behavioral: Text messaging plus nicotine replacement therapy
- Standard Care (Active Comparator): Advice to quit and brief discussion of tobacco use
  Interventions: Other: Standard Care at Lung Cancer Screening

INTERVENTIONS:
Behavioral: Text messaging plus nicotine replacement therapy — Brief advice to quit smoking prior to lung cancer screening (LCS), 8 weeks of gain-framed, LCS-tailored text messages, and nicotine replacement therapy.
  Arms: Treatment Arm
Other: Standard Care at Lung Cancer Screening — Brief advice to quit smoking prior to lung cancer screening
  Arms: Standard Care

SUMMARY:
The proposed study will test a medication plus text messaging intervention specifically designed for lung cancer screening patients. Half of the patients will receive standard of care, and half will receive the treatment intervention.

DETAILED DESCRIPTION:
Screening for lung cancer at earlier, more treatable stages has the potential to reduce mortality from the U.S.'s most deadly cancer. Annual lung cancer screening with low-dose computed tomography is now recommended for high risk individuals based on age and smoking history. This study will evaluate a smoking cessation intervention for lung cancer screening patients. We will evaluate quit rates after a standard intervention (brief counseling session at time of lung cancer screening) versus a dual nicotine replacement therapy (NRT) and gain-framed text messaging intervention.

ELIGIBILITY:
Inclusion:

1. 55 years or older
2. 30 pack year history of smoking
3. current smoker (defined as breath carbon monoxide>6ppm)
4. willing to be randomized
5. English speaking

Exclusion:

1. unstable psychiatric/medical conditions such as suicidal ideation, acute psychosis, severe alcohol dependence, substance abuse, or dementia
2. in the immediate (within 2 weeks) post myocardial infarction period
3. serious arrhythmias
4. unstable angina pectoris
5. hemodynamically or electrically unstable
6. currently taking part in any other tobacco treatment program or using cessation medication (i.e., taking NRT or other cessation medications, enrolled in the Quitline, in another drug study).

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alana Rojewski, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 participants were consented in to the study, but 7 withdrew before randomization.
Period: Overall Study
Arm/Group | Treatment Arm | Standard Care
Started | 21 | 20
Completed | 21 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 48 individuals were consented in to the study, but 7 withdrew before randomization and 1 withdrew after randomization. Those data are not included in baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Standard Care | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (6.1) | 63.4 (6.3) | 64.4 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 19 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 15 | 11 | 26
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: End of Treatment Abstinence Rates
Description: 7-day point prevalence abstinence
Time Frame: Week 8 (end of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Standard Care
Number analyzed (Participants) | 21 | 19
Participants | 3 | 0

2. Secondary Outcome: End of Study Abstinence Rates
Description: Effect size estimates at End of Study
Time Frame: 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Standard Care
Number analyzed (Participants) | 21 | 19
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the duration of the study (20 weeks)
Arm/Group | Treatment Arm | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03927989/Prot_SAP_000.pdf